CLINICAL TRIAL: NCT02798744
Title: SGLT-2 Inhibitor Empagliflozin Effects on Appetite and Weight Regulation: A Randomised Double-blind Placebo-controlled Trial (The SEESAW Study)
Brief Title: SGLT-2 Inhibitor Empagliflozin Effects on Appetite and Weight Regulation.
Acronym: SEESAW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: Loughborough University (Other); University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0526
Record Dates: First submitted 2016-02-10; First posted 2016-06-14 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Empagliflozin 25mg once daily (Experimental): Empagliflozin (Jardiance™) 25mg once daily (orally)
  Interventions: Drug: Empagliflozin
- Empagliflozin 25mg once daily + diet (Experimental): Empagliflozin (Jardiance™) 25mg once daily (orally) + energy restriction diet
  Interventions: Drug: Empagliflozin; Behavioral: Diet
- Placebo once daily (Placebo Comparator): Placebo once daily (orally)
  Interventions: Drug: Placebo
- Placebo once daily + diet (Active Comparator): Placebo once daily (orally) + energy restriction diet
  Interventions: Behavioral: Diet; Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — 25mg once daily to be taken orally for the duration of the study (24 weeks)
  Other Names: Jardiance
  Arms: Empagliflozin 25mg once daily; Empagliflozin 25mg once daily + diet
Behavioral: Diet — Daily energy restriction diet to be followed for the duration of the study (24 weeks)
  Other Names: Energy restriction diet
  Arms: Empagliflozin 25mg once daily + diet; Placebo once daily + diet
Drug: Placebo — Placebo once daily for the duration of the study (24 weeks)
  Arms: Placebo once daily; Placebo once daily + diet

SUMMARY:
The aim of this study is to investigate the cause for the discrepancy in predicted and observed weight loss with Empagliflozin (Jardiance™) by measuring appetite regulation.

Major secondary objectives are to determine the effects of Empagliflozin (Jardiance™) on energy expenditure and change in total body weight and body composition.

The primary outcome is change in appetite hormone concentrations (specifically total PYY) between baseline and 24 weeks: - this will be measured by sequential blood sampling during visits 1-5.

Secondary outcomes, which are exploratory, are effect on appetite hormones (ghrelin and GLP-1), appetite perceptions, total body weight and fat and fat free mass, energy expenditure, appetite perception, physical activity and blood and urine biochemical parameters after Empagliflozin (Jardiance™) treatment for 24 weeks.

The sample size for the study is 76 participants and the planned trial duration is 21 months, with participants receiving approximately 24 weeks of exposure to Empagliflozin (Jardiance™).

DETAILED DESCRIPTION:
Out of a family of six sodium glucose co-transporters, two have been extensively studied for therapeutic indications involving glucose reabsorption from the glomerular filtrate. Sodium glucose co-transporter-1 (SGLT-1), which is mainly found in both the renal tubule and enterocytes lining intestinal villi, transfers glucose across a concentration gradient resulting in glucose absorption from the gut and accounting for 10% of the glucose reabsorption from the renal tubules. Sodium glucose co-transporter-2 (SGLT-2), which is mostly found in the kidneys, is responsible for reabsorbing 90% of the glucose that is filtered by the renal tubules. Compared with healthy individuals, SGLT-2 is over-expressed and over-activated in those with type 2 diabetes.

SGLT-2 inhibitors are a new class of glucose-lowering drugs for the management of type 2 diabetes which reduce plasma glucose levels by increasing urinary glucose excretion (UGE) by up to 60-80g (240-320 kilo Calories) per day. SGLT-1 inhibitors and combined SGLT-1 and -2 inhibitors are currently in development.

Several SGLT-2 inhibitors are commercially available and licensed for use in the UK including dapagliflozin, canagliflozin and Empagliflozin (Jardiance™). They all lower glycated haemoglobin (HbA1c) effectively compared with placebo (mean difference vs. placebo -0.66% (95% Confidence Interval, -0.73% to -0.58%). They also result in weight loss of approximately 1.8kg compared with placebo and in combination with other oral hypoglycaemic medications. Some of this weight loss can be attributed to fluid loss due to osmotic diuresis from UGE. Weight is lost from both subcutaneous and visceral stores of adipose tissue.

Phase II studies have shown that the highly selective and potent SGLT-2 inhibitor Empagliflozin (Jardiance™) results in significant reductions in HbA1c level after 12 weeks of therapy compared with placebo (HbA1c 0.4-0.6% reduction with 5-25mg daily dose, p<0.0001) and reduction was similar to that seen with metformin. Weight loss of between 1.81-2.33kg was also achieved depending on Empagliflozin (Jardiance™) dose along with reduction in fasting plasma glucose (FPG). Similar improvements in HbA1c, weight and FPG have been seen in phase III trials with Empagliflozin (Jardiance™) both as monotherapy and in combination with metformin, sulphonylureas or insulin.

Empagliflozin (Jardiance™) is licensed in the UK for use in type 2 diabetes management. In this study, we will be using Empagliflozin (Jardiance™) according to its licensed indications and dosage. The commonest known side-effects include urinary tract and genital mycotic infections which are more frequent in women than men and generally mild in severity. Dehydration and postural hypotension may occur due to volume depletion and modest lowering of blood pressure. Increased urinary frequency may also occur. Increased risk of hypoglycaemia is observed when Empagliflozin (Jardiance™) is combined with sulphonylureas or insulin.

Weight loss from increased UGE and net energy loss with SGLT-2 inhibitors is less than expected as shown by studies in patients with type 2 diabetes. Endogenous glucose production is markedly increased with shifting of substrate utilisation from carbohydrate to lipid.

Up to 90g of glucose are excreted per day with Empagliflozin (Jardiance™) which equates to 360 kilo Calories per day lost by glycosuria. A 90 week study of patients with type 2 diabetes treated with Empagliflozin (Jardiance™) 25mg daily showed that average weight loss was 3.2±4.2kg representing a calorie deficit of 51 kilo Calories /day (interquartile range 112). This was 29%±41% of the expected loss of 11.3±3.1kg predicted by glycosuria of 206 kilo Calories per day using a validated mathematical model (http://bwsimulator.niddk.nih.gov). An increase in daily calorie intake of 269 kilo Calories /day [Inter Quartile Range 258] and daily energy expenditure appear to be the adaptive responses due to Empagliflozin (Jardiance™) therapy and the combination of SGLT-2 inhibitors and calorie restriction has been recommended by the authors of this study.

Appetite stimulation resulting in increased energy intake may be the underlying mechanism for this weight loss deficit. Furthermore, glucagon response is increased by SGLT-2 inhibition using Empagliflozin (Jardiance™) and dapagliflozin.

Appetite hormones such as peptide Y-Y (PYY) and ghrelin are important in the control of appetite and weight regulation. They are secreted from intestinal L cells which are found in the distal small intestine. Ghrelin, which stimulates hunger, has been shown to increase with weight loss and energy restriction diets. Glucagon-like peptide 1 (GLP-1) is another hormone which is involved in the regulation of appetite and satiety along with other glucose homeostatic effects.

There are no studies that have investigated the impact of SGLT-2 inhibitors on appetite hormones and effect on body composition. It is essential to understand these mechanisms in order to maximize the weight loss achievable with these agents. They may need to be combined with appropriate dietary measures such as energy restriction diets and weight-lowering or weight-neutral hypoglycaemic therapies for optimal clinical benefit. The aim of our study is to explore the relationship between appetite hormones and Empagliflozin (Jardiance™) in order to understand the underlying mechanisms for observed weight loss which does not equate with that predicted for these agents.

Primary Objective:

The aim of this study is to investigate the cause for the discrepancy in predicted and observed weight loss with Empagliflozin (Jardiance™) by measuring appetite regulation.

Secondary Objectives:

To determine the effects of Empagliflozin (Jardiance™) on resting energy expenditure and change in total body weight and body composition.

Study End Points:

The primary endpoint is effect on appetite hormones (specifically total PYY) with Empagliflozin (Jardiance™) after treatment for 24 weeks.

Secondary endpoints, which are exploratory, are effect on:

(i) Appetite hormones ghrelin and GLP-1 and appetite perception (ii) Total body weight and change in body composition (fat and fat free mass) (iii) Resting energy expenditure (iv) Physical activity (v) Change in blood and urine biochemical parameters.

This study is a randomised, double-blind placebo-controlled trial conducted over 24 weeks in male and postmenopausal female participants with type 2 diabetes on lifestyle control or stable metformin dose only to compare the effects of Empagliflozin (Jardiance™) on appetite and weight regulation compared with placebo and energy restriction diet.

Participants will be randomised to one of four arms at baseline:- (i) Empagliflozin (Jardiance™) 25mg once daily (ii) Empagliflozin (Jardiance™) 25mg once daily and energy restriction diet (iii) Placebo (iv) Placebo and energy restriction diet Participants will be stratified for age and BMI. STUDY CONDUCT Participant Withdrawal:- Each participant has the right to withdraw from the study at any time without needing to give a reason. The investigator may discontinue a participant from the study at any time if considered necessary. The reason for withdrawal will be recorded in the CRF and medical records. If the participant is withdrawn due to an adverse event, the investigator will arrange for follow-up visits or telephone calls until the adverse event has resolved or stabilised. The duration of safety follow-ups will be at least five half-lives of the study medication. The half-life of Empagliflozin (Jardiance™) is 12.4 hours, thus the duration of safety follow-ups will be rounded up to be at least 72 hours (or 3 days). The participant will be withdrawn from the study if they lose capacity and data collected up to that point will be used for analysis. As analysis will be on an intention-to-treat basis, there will be analysis of all data of participants receiving study medication (e.g. most safety analyses) and data will be admitted to the database even after the participant has withdrawn from the study.

Source Data:- Source documents are original documents, data, and records from which participants' CRF data will be obtained. These include, but are not limited to, hospital records (from which medical history and previous and concurrent medication will be summarised into the CRF), clinical and office charts, laboratory and pharmacy records, diaries, microfiches, radiographs, and correspondence. On all study-specific documents, other than the signed consent, the participant will be referred to by the study participant number/code only, and not by name.

Drug Management:- The licensed product Empagliflozin (Jardiance™) will be handled according to the University Hospitals of Leicester pharmacy in-house protocols.

Compliance with Study Treatment:- The participants will be instructed to return all unused or part-used medication and packaging from used medication at each visit. The Investigator may withdraw the participants if they consider dose compliance is unsatisfactory.

Concomitant Medication:- Throughout the study, Investigators will be able to prescribe any concomitant medications or treatments deemed necessary to provide adequate supportive care except for those listed in the exclusion criteria. If these are required, the participant will be withdrawn. Any medication, other than the study medication taken during the study will be recorded in the CRF. Contraindicated medications during the study will include any other glucose-lowering therapies apart from metformin. Loop diuretic therapy will also be contraindicated. As study drug Empagliflozin (Jardiance™), placebo and metformin do not cause hypoglycaemia, participants will not be expected to perform home blood glucose monitoring during the study.

SAFETY REPORTING Expected Serious Adverse Events/Reactions (SAE):- The most common adverse events seen with Empagliflozin (Jardiance™) are urinary tract and mycotic fungal infections (e.g. balanitis) and volume depletion leading to dehydration, postural hypotension and dizziness. If these events lead to hospitalisation of the participant, they will require immediate reporting to the study team. Otherwise, they will be treated as an AE and need reporting to the study team within 2 working days.

Abnormalities of renal and liver function will also be closely monitored as part of the usual study visits and any significant clinical deterioration in renal and/or liver function will be reported as an SAE. A serious deterioration in renal function to be classified as an SAE will be a reduction in eGFR to less than 30ml/min/1.73m2. A serious deterioration in liver function will be classified as an SAE if ALT (Alanine aminotransferase) or AST (Aspartate aminotransferase) is 3 x greater than the upper limit of normal.

Ketoacidosis and Diabetic Ketoacidosis (DKA) have recently been reported as a possible serious SAE occurring with SGLT-2 inhibitor use by the US Food and Drugs Administration. Participants will be closely monitored for the development of this SAE and will be advised to seek medical attention immediately if they experience symptoms such as difficulty breathing, nausea, vomiting, abdominal pain, confusion, unusual fatigue or sleepiness, anorexia, excessive thirst, dehydration, low food intake, weight loss, infection, poor control of diabetes, and/or only moderately increased glucose levels.

In patients where DKA is suspected or diagnosed, treatment with SGLT-2 inhibitors will be discontinued immediately. Restarting SGLT-2 inhibitor treatment in patients with previous DKA while on SGLT-2 inhibitor treatment is not recommended unless another clear precipitating factor is identified and resolved. Treatment will also be interrupted in patients who are hospitalised for major surgical procedures or acute medical illnesses. In both cases, treatment with SGLT-2 inhibitors may be restarted once the patient's condition has stabilised and only once the necessary safety assessments have been performed. The decision to stop or interrupt and subsequently re-start the study treatment Empagliflozin (Jardiance™) will be documented in the participant's medical notes. Any decisions regarding the withdrawal of participants from the study will be made by the study clinician and Principal Investigator.

Suspected Unexpected Serious Adverse Reactions (SUSAR) A serious adverse reaction, the nature or severity of which is not consistent with the Summary of Product Characteristics for Empagliflozin (Jardiance™) will be reported as a SUSAR.

Adverse Events of Special Interests (AESI) Adverse Events of Special Interests (AESI)

* Decreased renal function: creatinine value shows a ≥ 2 fold increase from baseline and is above ULN
* Hepatic injury defined by the following alterations of liver parameters after randomization at visit 1:-

  * Elevation of AST and/or ALT≥3 fold ULN combined with an elevation of total bilirubin≥2 fold ULN measured in the same blood draw sample
  * Isolated elevation of AST and/or ALT≥5 fold ULN irrespective of any bilirubin elevation
* Diabetic Ketoacidosis (DKA) o DKA is defined by the diagnostic criteria in the table below, and as defined by the American Diabetes Association (ADA).

Investigators should note that not all criteria in Table 2 (below) need to apply for the diagnosis of DKA, and clinical judgment should also be taken into consideration. Due to its mechanism of action, Empagliflozin (Jardiance™) may potentially modify the clinical presentation of DKA which may occur at lower plasma glucose levels.

If any AESIs occur they will be reported to the Sponsor and Boehringer Ingelheim using the same procedure as reporting Serious Adverse Events (SAEs).

Reporting Procedures for Serious Adverse Events:- All SAEs will be reported internally to the Sponsor within one working day (24 hours) of discovery or notification of the event. The SAE will be reported using appropriate forms and the immediate report will be made in writing and shall be followed by a detailed written report of the event. Additional information can be provided if requested to the Sponsor and main Research Ethics Committee (REC) (e.g. in the event of a death). The Principal Investigator or another delegated physician is responsible for the review and sign off of the SAE, or in their absence, another member of the team (in order to avoid a delay).

The Sponsor will perform an initial check of the information and ensure that it is reviewed at the next R&D management meeting. All SAE information must be recorded on an SAE form and sent to the Sponsor. Additional information received for a case (follow-up or corrections to the original case) needs to be detailed on a new SAE form and sent to the Sponsor.

The Sponsor will report all SUSARs to the MHRA and the REC concerned. Fatal or life-threatening SUSARs must be reported within 7 days and all other SUSARs within 15 days. The Chief Investigator will inform all investigators concerned of relevant information about SUSARs that could adversely affect the safety of participants. The Sponsor will use the Summary of Product Characteristics (SmPC) as the Reference Safety Information (RSI) when determining the expectedness of any untoward medical occurrences and thus SAE/SUSAR reporting.

In addition to the expedited reporting above, the Chief Investigator will submit once a year throughout the clinical study or on request a Developmental Safety Update Report (DSUR) to the MHRA and REC. The PI will inform all investigators concerned of relevant information about SUSARs that could adversely affect the safety of participants.

STATISTICS Description of Statistical Methods:- Participants recruited to the study will be compared within and by treatment group. For the latter, each active treatment arm, whether medication, medication and energy restriction diet or placebo and energy restriction diet, will be compared against the placebo only arm. Baseline variables will be presented by arm using N (%) for categorical variables and mean (standard deviation) or median (interquartile range) as appropriate, for continuous variables.

The primary outcome is change in appetite hormones from baseline to week 24 within and between treatment groups. AUC values for appetite hormone measurements at baseline and 24 weeks will be calculated using the trapezoidal rule. Paired t-tests or equivalent non-parametric tests will be used to analyse the change in appetite hormones within individual treatment groups. One way analysis of variance will be used to calculate mean changes in AUC from baseline to 24 weeks by treatment group. Adjusted treatment effects will be calculated via linear regression analysis or similarly appropriate methods, to compare each treatment against placebo. Models will include a categorical treatment variable and will be adjusted for stratification factors; age and BMI as well as baseline AUC value. Changes in appetite hormones from baseline to weeks 2, 6 and 12 will also be analysed using the same methods; however will represent hypothesis generating analyses only. Similarly, overall changes in appetite hormones over time will be analysed using multilevel models, adjusted for stratification factors.

The analysis for the primary outcome will be repeated for secondary endpoints; changes in resting energy expenditure, weight and body composition, physical activity and biochemical parameters from baseline.

All analyses of outcome data will be carried out on a complete case basis, so only those patients with complete data will be included in the analysis. Intention to treat and per protocol analyses will be carried out as sensitivity analyses, using multiple imputation and including only those who remain on their treatment regimen for the duration of the study, respectively.

The Number of Participants:- The power calculation is based on the primary outcome of change in appetite hormones and a standard deviation of area under the curve of 96.2pg/ml of total PYY based on a study looking at the influence of resistance and aerobic exercise on hunger and circulating levels of total PYY in healthy males. To detect a minimum clinically significant difference of 120pg/ml in area under the curve of total PYY between groups, we will require 15 participants in each of the four arms with 80% power and 2-sided alpha of 1.7%. This will allow three comparisons between arms. To account for up to 20% dropout, 19 participants will be required in each arm; therefore 76 participants will be recruited in total.

The Level of Statistical Significance:- Statistical significance will be taken at the level of p<0.05. QUALITY CONTROL AND QUALITY ASSURANCE PROCEDURES The study will be conducted in accordance with the current approved protocol, International Conference on Harmonisation Good Clinical Practice, relevant regulations and standard operating procedures (SOPs).

Regular monitoring will be performed according to International Conference on Harmonisation Good Clinical Practice. Data will be evaluated for compliance with the protocol and accuracy in relation to source documents. Following written standard operating procedures, the monitors will verify that the clinical trial is conducted and data are generated, documented and reported in compliance with the protocol, Good Clinical Practice and the applicable regulatory requirements.

STUDY GOVERNANCE The study will be conducted in accordance with the Research Governance Framework for Health and Social Care, ICH GCP and the Data Protection Act. The Sponsor responsible for checking research governance arrangements will be the University of Leicester. A Trial Steering Committee (TSC), Data Safety Monitoring Committee (DSMC) and Project Management Committee (PMC) will be set up to support the running of the study.

ELIGIBILITY:
Inclusion Criteria

1. Male and postmenopausal female participants aged between 30-75 years of age inclusive
2. Type 2 diabetes on diet and lifestyle control or stable dose of metformin only for at least 3 months
3. Stable weight (less than 5% change in body weight in last 3 months) - determined by self-reporting or documentation in clinical records
4. HbA1c 48-86mmol/mol (6.0 - 10%)
5. eGFR≥60ml/min/1.73m2
6. BMI ≥ 25kg/m2
7. Able and willing to give informed consent
8. Able to understand English

Exclusion Criteria

1. Females who are not postmenopausal (as menstrual cycle can affect appetite hormone concentrations) which is defined as "2 years post last menstrual period <50 years of age or 1 year post last menstrual period >50 years of age."
2. Type 2 diabetes on any other glucose lowering treatment except metformin
3. Patients with Type 1 diabetes
4. Patients on loop diuretics
5. Age <30 years and >75 years
6. BMI <25kg/m2
7. Not able to give informed consent
8. Not able to understand English
9. Moderate to severe renal impairment (eGFR<60ml/min/1.73m2)
10. Unstable diabetes i.e. HbA1c >86mmol/mol (10%), recent hospital admission with diabetic emergency in last 3 months
11. Patients with familial renal glycosuria
12. Patients with recurrent balanitis, vaginal or urinary tract infections
13. Shift workers
14. Patients who have participated in another study of an investigational medicinal product in the last 3 months
15. Active malignancy
16. Serious illness with a life-expectancy of less than 1 year
17. Hypersensitivity to Empagliflozin (Jardiance™) or to any of the excipients
18. Patients with latent autoimmune diabetes in adults (LADA)
19. Patients with a history of chronic pancreatitis
20. Evidence of conditions that lead to restricted food intake or severe dehydration
21. Patients with a history of excessive alcohol consumption
22. Patients on a severely calorie restricted diet (i.e., ≤800 calories per day)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Total PYY at 24 weeks | Baseline and 24 weeks
  The effect of Empagliflozin on appetite hormone 'Total PYY' concentration between baseline and 24 weeks. Measured by sequential blood sampling at study visits 1-5.

SECONDARY OUTCOMES:
Change from baseline in Ghrelin at 24 weeks | Baseline and 24 weeks
  Change in appetite hormone 'Ghrelin' concentration from baseline to 24 weeks. Measured by blood sampling at study visits 1-5.
Change from baseline in GLP-1 to 24 weeks | Baseline and 24 weeks
  Change in appetite hormone 'GLP-1' concentration from baseline to 24 weeks. Measured by blood sampling at study visits 1-5.
Change from baseline in appetite perceptions to 24 weeks | Baseline and 24 weeks
  Change in appetite perceptions from baseline to 24 weeks. Measured by questionnaires visits 1 -5.
Change in Weight (kg) from baseline to 24 weeks | Baseline and 24 weeks
  Change in weight (kg) from baseline to study end and between groups. This will be measured at visits 1 - 5.
Change in Body composition from baseline to 24 weeks | Baseline and 24 weeks
  Change in body composition from baseline to study end and between groups. This will be measured by Dual Energy X-Ray Absorptiometry (DEXA) scanning at visits 1 and 5.
Change in resting energy expenditure from baseline to 24 weeks | Baseline and 24 weeks
  Change in resting energy expenditure from baseline to study end and between groups. This will be measured by indirect calorimetry at visits 1-5.
Change in objectively measured Physical Activity from baseline to 24 weeks using activity monitors | Baseline and 24 weeks
  Change in physical activity from baseline to study end and between groups. This will be measured using physical activity monitors at visits 0, 3, 4 and 5.
Change in subjectively measured Physical Activity from baseline to 24 weeks using the International Physical Activity Questionnaire (IPAQ) | Baseline and 24 weeks
  Change in physical activity from baseline to study end and between groups. This will be measured using the international physical activity questionnaire at visits 1 - 5.
Change from baseline urine glucose excretion to 24 weeks. | Baseline and 24 weeks
  Change in urine glucose excretion to study end and between groups. This will be measured using urine sampling at visits 1-5.
Change from baseline in blood appetite hormones to 24 weeks | Baseline and 24 weeks
  Change in in baseline blood appetite hormones to 24 weeks between groups. This will be measured using blood sampling at visits 1-5.
Change from baseline in HbA1c to 24 weeks | Baseline and 24 weeks
  Change in in baseline HbA1c to 24 weeks between groups. This will be measured using blood sampling at visits 1-5.
Change from baseline in inflammatory markers to 24 weeks | Baseline and 24 weeks
  Change in in baseline inflammatory markers to 24 weeks between groups. This will be measured using blood sampling at visits 1-5.
Change from baseline in renal functioning to 24 weeks | Baseline and 24 weeks
  Change in in baseline renal functioning to 24 weeks between groups. This will be measured using blood sampling at visits 1-5.
Change from baseline in liver functioning to 24 weeks | Baseline and 24 weeks
  Change in in baseline liver functioning to 24 weeks between groups. This will be measured using blood sampling at visits 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J Davies, MBBS MD FRCP, Principal Investigator — University of Leicester
Locations (1):
- Leicester Diabetes Centre, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey CJ. Renal glucose reabsorption inhibitors to treat diabetes. Trends Pharmacol Sci. 2011 Feb;32(2):63-71. doi: 10.1016/j.tips.2010.11.011. Epub 2011 Jan 4. PMID 21211857
- [Background] Bailey CJ. SGLT2 inhibitors:Glucuretic treatment for type 2 diabetes. British Journal of Diabetes and Vascular Disease. 2010;10:193-199
- [Background] Hasan FM, Alsahli M, Gerich JE. SGLT2 inhibitors in the treatment of type 2 diabetes. Diabetes Res Clin Pract. 2014 Jun;104(3):297-322. doi: 10.1016/j.diabres.2014.02.014. Epub 2014 Mar 11. PMID 24735709
- [Background] Bolinder J, Ljunggren O, Kullberg J, Johansson L, Wilding J, Langkilde AM, Sugg J, Parikh S. Effects of dapagliflozin on body weight, total fat mass, and regional adipose tissue distribution in patients with type 2 diabetes mellitus with inadequate glycemic control on metformin. J Clin Endocrinol Metab. 2012 Mar;97(3):1020-31. doi: 10.1210/jc.2011-2260. Epub 2012 Jan 11. PMID 22238392
- [Background] Broom DR, Batterham RL, King JA, Stensel DJ. Influence of resistance and aerobic exercise on hunger, circulating levels of acylated ghrelin, and peptide YY in healthy males. Am J Physiol Regul Integr Comp Physiol. 2009 Jan;296(1):R29-35. doi: 10.1152/ajpregu.90706.2008. Epub 2008 Nov 5. PMID 18987287
- [Background] Ferrannini E, Seman L, Seewaldt-Becker E, Hantel S, Pinnetti S, Woerle HJ. A Phase IIb, randomized, placebo-controlled study of the SGLT2 inhibitor empagliflozin in patients with type 2 diabetes. Diabetes Obes Metab. 2013 Aug;15(8):721-8. doi: 10.1111/dom.12081. Epub 2013 Mar 4. PMID 23398530
- [Background] Ferrannini E, Muscelli E, Frascerra S, Baldi S, Mari A, Heise T, Broedl UC, Woerle HJ. Metabolic response to sodium-glucose cotransporter 2 inhibition in type 2 diabetic patients. J Clin Invest. 2014 Feb;124(2):499-508. doi: 10.1172/JCI72227. Epub 2014 Jan 27. PMID 24463454
- [Background] Ferrannini G, Hach T, Crowe S, Sanghvi A, Hall KD, Ferrannini E. Energy Balance After Sodium-Glucose Cotransporter 2 Inhibition. Diabetes Care. 2015 Sep;38(9):1730-5. doi: 10.2337/dc15-0355. Epub 2015 Jul 15. PMID 26180105
- [Background] Haring HU, Merker L, Seewaldt-Becker E, Weimer M, Meinicke T, Woerle HJ, Broedl UC; EMPA-REG METSU Trial Investigators. Empagliflozin as add-on to metformin plus sulfonylurea in patients with type 2 diabetes: a 24-week, randomized, double-blind, placebo-controlled trial. Diabetes Care. 2013 Nov;36(11):3396-404. doi: 10.2337/dc12-2673. Epub 2013 Aug 20. PMID 23963895
- [Background] Haring HU, Merker L, Seewaldt-Becker E, Weimer M, Meinicke T, Broedl UC, Woerle HJ; EMPA-REG MET Trial Investigators. Empagliflozin as add-on to metformin in patients with type 2 diabetes: a 24-week, randomized, double-blind, placebo-controlled trial. Diabetes Care. 2014 Jun;37(6):1650-9. doi: 10.2337/dc13-2105. Epub 2014 Apr 10. PMID 24722494
- [Background] Kovacs CS, Seshiah V, Swallow R, Jones R, Rattunde H, Woerle HJ, Broedl UC; EMPA-REG PIO trial investigators. Empagliflozin improves glycaemic and weight control as add-on therapy to pioglitazone or pioglitazone plus metformin in patients with type 2 diabetes: a 24-week, randomized, placebo-controlled trial. Diabetes Obes Metab. 2014 Feb;16(2):147-58. doi: 10.1111/dom.12188. Epub 2013 Aug 22. PMID 23906415
- [Background] Madsbad S. The role of glucagon-like peptide-1 impairment in obesity and potential therapeutic implications. Diabetes Obes Metab. 2014 Jan;16(1):9-21. doi: 10.1111/dom.12119. Epub 2013 May 26. PMID 23617798
- [Background] Merovci A, Solis-Herrera C, Daniele G, Eldor R, Fiorentino TV, Tripathy D, Xiong J, Perez Z, Norton L, Abdul-Ghani MA, DeFronzo RA. Dapagliflozin improves muscle insulin sensitivity but enhances endogenous glucose production. J Clin Invest. 2014 Feb;124(2):509-14. doi: 10.1172/JCI70704. Epub 2014 Jan 27. PMID 24463448
- [Background] Mifflin MD, St Jeor ST, Hill LA, Scott BJ, Daugherty SA, Koh YO. A new predictive equation for resting energy expenditure in healthy individuals. Am J Clin Nutr. 1990 Feb;51(2):241-7. doi: 10.1093/ajcn/51.2.241. PMID 2305711
- [Background] Rahmoune H, Thompson PW, Ward JM, Smith CD, Hong G, Brown J. Glucose transporters in human renal proximal tubular cells isolated from the urine of patients with non-insulin-dependent diabetes. Diabetes. 2005 Dec;54(12):3427-34. doi: 10.2337/diabetes.54.12.3427. PMID 16306358
- [Background] Ridderstrale M, Andersen KR, Zeller C, Kim G, Woerle HJ, Broedl UC; EMPA-REG H2H-SU trial investigators. Comparison of empagliflozin and glimepiride as add-on to metformin in patients with type 2 diabetes: a 104-week randomised, active-controlled, double-blind, phase 3 trial. Lancet Diabetes Endocrinol. 2014 Sep;2(9):691-700. doi: 10.1016/S2213-8587(14)70120-2. Epub 2014 Jun 16. PMID 24948511
- [Background] Roden M, Weng J, Eilbracht J, Delafont B, Kim G, Woerle HJ, Broedl UC; EMPA-REG MONO trial investigators. Empagliflozin monotherapy with sitagliptin as an active comparator in patients with type 2 diabetes: a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Diabetes Endocrinol. 2013 Nov;1(3):208-19. doi: 10.1016/S2213-8587(13)70084-6. Epub 2013 Sep 9. PMID 24622369
- [Background] Rosenstock J, Jelaska A, Frappin G, Salsali A, Kim G, Woerle HJ, Broedl UC; EMPA-REG MDI Trial Investigators. Improved glucose control with weight loss, lower insulin doses, and no increased hypoglycemia with empagliflozin added to titrated multiple daily injections of insulin in obese inadequately controlled type 2 diabetes. Diabetes Care. 2014 Jul;37(7):1815-23. doi: 10.2337/dc13-3055. Epub 2014 Jun 14. PMID 24929430
- [Background] Sumithran P, Prendergast LA, Delbridge E, Purcell K, Shulkes A, Kriketos A, Proietto J. Long-term persistence of hormonal adaptations to weight loss. N Engl J Med. 2011 Oct 27;365(17):1597-604. doi: 10.1056/NEJMoa1105816. PMID 22029981
- [Background] Tahrani AA, Barnett AH, Bailey CJ. SGLT inhibitors in management of diabetes. Lancet Diabetes Endocrinol. 2013 Oct;1(2):140-51. doi: 10.1016/S2213-8587(13)70050-0. Epub 2013 Aug 13. PMID 24622320
- [Background] Vasilakou D, Karagiannis T, Athanasiadou E, Mainou M, Liakos A, Bekiari E, Sarigianni M, Matthews DR, Tsapas A. Sodium-glucose cotransporter 2 inhibitors for type 2 diabetes: a systematic review and meta-analysis. Ann Intern Med. 2013 Aug 20;159(4):262-74. doi: 10.7326/0003-4819-159-4-201308200-00007. PMID 24026259
- [Derived] Sargeant JA, King JA, Yates T, Redman EL, Bodicoat DH, Chatterjee S, Edwardson CL, Gray LJ, Poulin B, Waheed G, Waller HL, Webb DR, Willis SA, Wilding JPH, Khunti K, Stensel DJ, Davies MJ. The effects of empagliflozin, dietary energy restriction, or both on appetite-regulatory gut peptides in individuals with type 2 diabetes and overweight or obesity: The SEESAW randomized, double-blind, placebo-controlled trial. Diabetes Obes Metab. 2022 Aug;24(8):1509-1521. doi: 10.1111/dom.14721. Epub 2022 May 13. PMID 35441435